CLINICAL TRIAL: NCT02672176
Title: Patient and Provider Engagement and Empowerment Through Technology (P2E2T2) Program to Improve Health in Diabetes
Brief Title: Improving Health in Diabetes Project
Acronym: P2E2T2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 820612
Record Dates: First submitted 2016-01-20; First posted 2016-02-03 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; Motivational Interviewing; Mobile Health Technology; Patient-generated Health Data (PGHD)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care-Chronic Disease Management (Sham Comparator): Usual Care through Chronic Disease Management: The role of the care coordinator is to assess needs of the patient and coordinate healthcare referrals and appointments for the patient, facilitate communication among members of the healthcare team, identify health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient. Contact is variable and conducted on a case by case basis.
  Interventions: Behavioral: Usual Care
- P2E2T2 Program (Active Comparator): The P2E2T2 intervention group will receive Nurse Health Coaching using MI, an approach designed to elicit and support behavioral changes and improve self-efficacy (2, 3). Nurses delivering the intervention will have completed the Health Science Institutes Registered Health Coach (RHC) training program (www.healthsciences.org).
  Interventions: Behavioral: P2E2T2 Program

INTERVENTIONS:
Behavioral: Usual Care — This program is a well-established program within the UC Davis Health System, providing care coordination to individuals with chronic conditions. Patients can self-refer or are referred by their providers for this service. The role of the care coordinator is to assess needs of the patient and coordinate healthcare referrals and appointments for the patient, facilitate communication among members of the healthcare team, identify health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient. Contact is variable and conducted on a case by case basis.
  Arms: Usual Care-Chronic Disease Management
Behavioral: P2E2T2 Program — The P2E2T2 intervention group will receive Nurse Health Coaching using MI, an approach designed to elicit and support behavioral changes and improve self-efficacy (18-21). Nurses delivering the intervention will have completed the Health Science Institutes Registered Health Coach (RHC) training program (www.healthsciences.org). The intervention protocol is as follows:
  Arms: P2E2T2 Program

SUMMARY:
The overall goal of this proposal is to enhance the supports and resources available to patients with diabetes to assist them to achieve their health goals. The investigators will evaluate an innovative program that uses nurse health coaching, motivational interviewing techniques, wireless sensors and mobile health (mHealth) technology. In this program, patients will receive timely, tailored nurse coaching feedback to facilitate behavior change using mHealth technology, thus bridging bidirectional exchange of meaningful information among patient, nurse coach and provider. The investigators will conduct a randomized controlled trial among patients receiving chronic disease management at the University of California Davis(UC Davis) Primary Care Network. The patients who are eligible for inclusion in the study will be randomized to one of two arms of the trial: 1) Usual care (Care Coordination) administered by UC Davis Health Management and Education; or 2) the Patient and Provider Engagement and Empowerment through Technology (P2E2T2) Program to Improve Health in Diabetes. The hypothesis is that patients in the P2E2T2 arm of the study will be more engaged in identifying and achieving health goals related to their diabetes and will achieve better health outcomes compared to patients receiving usual care.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a growing public health problem highly amenable to prevention and health promotion interventions. Over 26 million people are diagnosed with diabetes, and an estimated 79 million people have pre-diabetes (1). Physical inactivity, poor eating habits, obesity and smoking are common risk factors for multiple chronic diseases, including DM, and are associated with premature deaths in the United States (2). Traditional interventions for diabetes emphasize education and typically do not address patient-generated health data (3). Motivational interviewing (MI) is a counseling tool to improve self-efficacy and support behavioral changes that has been used successfully in treatment of addictions and chronic conditions including diabetes (4-6). MI focuses on enhancing goal-setting skills by encouraging focus on manageable steps to improve overall health, establishing reasonable goals, and managing barriers and obstacles to goal attainment. Mobile health (mHealth) technology can be used to allow bi-directional, timely communication of data and tailored feedback between the patient and health care team; thus mHealth has the potential to change an individual' health behavior and prevent factors that lead to disease (7). This proposal tests the effectiveness of nurse coaches and the mHealth platform as resources to patients. Specifically, the investigators will test a mobile technology-enabled nurse coaching intervention as a means to engage and empower patients to set their own personal goals to address lifestyle and behavioral changes to better manage their diabetes and comorbidities. The addition of a wireless sensing wearable device to monitor participant activities (physical activity, energy expenditure and sleep quality) will allow the investigators to perform meaningful analysis of patient-generated health data and provide tailored feedback to motivate the patient to reach personal goals. The investigators will achieve this project through the following Specific Aims:

Specific Aim 1: To evaluate the effectiveness of the P2E2T2 program on diabetes management as measured by the following outcomes: 1) quality of life (QOL); 2) self-efficacy; 3) readiness to change; and 4) clinically relevant outcomes.

This study is a randomized, controlled trial with two groups: 1) Usual care (Care Coordination); and 2) the Patient and Provider Engagement and Empowerment Through Technology (P2E2T2) program - nurse coaching paired with mobile sensor technology to provide targeted feedback of patient-generated, real-world community physical activity and sleep quality data to the nurse coach, participants, and primary care providers to improve self-management of diabetes. Participants will be recruited from the UC Davis Primary Care Clinics network. After enrollment in the study, those randomized to receive the intervention will interact with their nurse coach through mobile technologies by telephone, or by text/e-mail through the secure mHealth dashboard platform established for communication and transfer of data. The investigators expect to enroll at least 150 patients in each of the intervention and control arms. This sample size will be sufficient to detect differences between the two groups. Even under the conservative assumption that design effects and dropout rates may result in a reduced sample size of 100 per treatment group, the study will still have at least 80% power to detect the specified clinically important effect size. Based on a previous study of nurse coaching using MI to improve disease self-management (8), the investigators found improvement in self-efficacy scores significantly higher in the intervention group compared to the control group. Data will be collected from participants at three time points: 1) baseline data at time of recruitment; 2) 3 months (coinciding with the completion of the intervention); and 3) 9 months (selected to assess sustained effects of the intervention (6 months after intervention ended)). At baseline, in addition to outcomes, all participants will complete a demographic survey which will include age, gender, race/ethnicity, education level, income level and insurance type and health history using the Charlson Comorbidity Index which includes common chronic conditions. All data for the study will be collected by the research coordinator and entered into the REDCap (Research Electronic Data Capture) system housed in the servers managed by UC Davis Clinical and Translational Science Center (CTSC) (9).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Diagnosis of Diabetes Mellitus (type 2)
3. Receiving care at one of the UC Davis Primary Care participating clinics (hospital-based Primary Care Clinic, the Folsom Primary Care Clinic)
4. Able to read, write, and speak English
5. Has access to a telephone and computing device
6. Has had experience with use of a mobile smartphone & applications
7. HgbA1C over 6.5%

Exclusion Criteria:

1. Does not have Diabetes Mellitus
2. Primary language is not English
3. Pregnant women
4. Those that not have access to a telephone or computing device
5. Has a HgbA1C value under 6.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Young, Principal Investigator — UC Davis
Locations (1):
- School of Nursing, University of California, Davis and UC Davis Health System, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Young HM, Miyamoto S, Dharmar M, Tang-Feldman Y. Nurse Coaching and Mobile Health Compared With Usual Care to Improve Diabetes Self-Efficacy for Persons With Type 2 Diabetes: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Mar 2;8(3):e16665. doi: 10.2196/16665. PMID 32130184
- [Derived] Miyamoto S, Dharmar M, Fazio S, Tang-Feldman Y, Young HM. mHealth Technology and Nurse Health Coaching to Improve Health in Diabetes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Feb 15;7(2):e45. doi: 10.2196/resprot.9168. PMID 29449200
- [Derived] Broadbent E, Garrett J, Jepsen N, Li Ogilvie V, Ahn HS, Robinson H, Peri K, Kerse N, Rouse P, Pillai A, MacDonald B. Using Robots at Home to Support Patients With Chronic Obstructive Pulmonary Disease: Pilot Randomized Controlled Trial. J Med Internet Res. 2018 Feb 13;20(2):e45. doi: 10.2196/jmir.8640. PMID 29439942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from three Primary Care Clinics at UC Davis Health
Groups:
- Usual Care-Chronic Disease Management: Usual Care through Chronic Disease Management: The role of the care coordinator is to assess needs of the patient and coordinate healthcare referrals/ appointments for the patient, facilitate communication among the healthcare team, identify health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient. Contact is variable and conducted on a case by case basis.
  Usual Care: This program is a well-established program within UC Davis Health, providing care coordination to individuals with chronic conditions. Patients can self-refer or are referred by their providers for this service. The care coordinator assesses the needs of the patient and coordinates healthcare referrals and appointments, facilitates communication among the healthcare team, identifies health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient.
- P2E2T2 Program: The P2E2T2 intervention group will receive Nurse Health Coaching using MI, an approach designed to elicit and support behavioral changes and improve self-efficacy (2, 3). Nurses delivering the intervention will have completed the Health Science Institutes Registered Health Coach (RHC) training program (www.healthsciences.org).
  P2E2T2 Program: The P2E2T2 intervention group will receive Nurse Health Coaching using motivational interviewing (MI), an approach designed to elicit and support behavioral changes and improve self-efficacy (18-21). Nurses delivering the intervention will have completed the Health Science Institutes Registered Health Coach (RHC) training program (www.healthsciences.org). The intervention protocol is as follows:
Period: Overall Study
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Started | 161 | 158
Completed | 155 | 132
Not Completed | 6 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program | Total
Number analyzed (Participants) | 155 | 132 | 287
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 89 | 192
  >=65 years | 52 | 43 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.16 (11.69) | 59.59 (11.17) | 59.36 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Three participants declined to indicate gender (1 participant in the intervention group and 2 in the control group)
  Participants
    Gender: number analyzed (Participants) | 154 | 130 | 284
    Gender: Female | 73 | 62 | 135
    Gender: Male | 81 | 68 | 149
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 16 | 11 | 27
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 18 | 19 | 37
  White | 96 | 76 | 172
  More than one race | 10 | 8 | 18
  Unknown or Not Reported | 12 | 13 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 155 | 132 | 287
Diabetes self-efficacy [Mean (Standard Deviation); unit: units on a scale] — Diabetes Empowerment Scale (DES)-Short Form - This eight-item instrument measures diabetes-related psychosocial self-efficacy using a 5-point Likert scale with raw scores ranging from 8 to 40. Total score is the sum of the eight questions divided by the number of items in the survey (range is 1 to 8), with higher scores indicating greater self-efficacy. A 0.25 point difference in this score is equivalent to a shift of at least one point in two questions in the DES tool; in other words, they have improved their confidence in engaging in self-management behavior in two areas.
  units on a scale | 3.66 (.89) | 3.67 (.83) | 3.66 (.85)

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Self-efficacy Measured Using the Diabetes Empowerment Scale Short Form (DES-SF)- Scores at Baseline
Description: Diabetes self-efficacy (Diabetes Empowerment Scale (DES)-Short Form) (http://diabetesresearch.med.umich.edu/Tools_SurveyInstruments.php). This eight-item survey instrument is derived from the 37 item DES survey, measuring diabetes-related psychosocial self-efficacy. The scale uses a 5-point Likert scale with raw scores on the scale ranging from 8 to 40. Total score is calculated as the sum of the eight questions divided by the number of items in the survey (range is 1 to 8), with higher scores indicating greater self-efficacy. The tool is a valid and reliable measure of overall diabetes-related psychosocial self-efficacy with an alpha of 0.84. Concurrent validity was established with attitudes about having diabetes, understanding diabetes and improved A1C scores. A 0.25 point difference in this score is equivalent to a shift of at least one point in two questions in the DES tool; in other words, they have improved their confidence in engaging in self-management behavior in two areas
Time Frame: Baseline
Population: Diabetes self-efficacy at baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 155 | 132
Units on a scale | 3.66 (0.89) | 3.67 (0.83)
Statistical Analysis 1: Comparison: Usual Care-Chronic Disease Management vs P2E2T2 Program; Test type: Equivalence — Information included in Statistical Analysis; p = 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Diabetes Self-Efficacy Measured Using the Diabetes Empowerment Scale Short Form (DES-SF)
Description: as for outcome 1
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usual Care-Chronic Disease Management: Usual Care through Chronic Disease Management: The role of the care coordinator is to assess needs of the patient and coordinate healthcare referrals and appointments for the patient, facilitate communication among members of the healthcare team, identify health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient. Contact is variable and conducted on a case by case basis.
  Usual Care: This program is a well-established program within the UC Davis Health System, providing care coordination to individuals with chronic conditions. Patients can self-refer or are referred by their providers for this service. The role of the care coordinator is to assess needs of the patient and coordinate healthcare referrals and appointments for the patient, facilitate communication among members of the healthcare team, identify health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient.
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 153 | 132
units on a scale | 3.71 (0.86) | 4.05 (0.69)
Statistical Analysis 1: Comparison: Usual Care-Chronic Disease Management vs P2E2T2 Program; Test type: Equivalence — See Statistical Analysis; p = 0.05, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Diabetes Self-Efficacy Measured Using the Diabetes Empowerment Scale Short Form (DES-SF)- Scores at 9-months
Description: as for outcome 1
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 149 | 131
units on a scale | 3.95 (0.97) | 3.97 (0.91)
Statistical Analysis 1: Comparison: Usual Care-Chronic Disease Management vs P2E2T2 Program; Test type: Equivalence — See Statistical Analysis; p = 0.05, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Depression Severity Measured by PHQ-9
Description: Depressive symptoms were measured with the PHQ-9. This is a 9-question instrument commonly administered to patients in a primary care setting to screen for the presence and severity of depression. The sum total of the responses ranges from 0 to 27. The total score determines the level of depressive symptoms. Higher scores indicate more depressive symptoms. In general, a score of 10 or above is suggestive of the presence of depression. This instrument has demonstrated validity and reliability with an alpha of 0.89 when evaluated in 3000 primary care patients.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 155 | 132
units on a scale | 5.36 (4.64) | 5.00 (4.99)
Statistical Analysis 1: Comparison: Usual Care-Chronic Disease Management vs P2E2T2 Program; Test type: Equivalence — See Statistical Analysis; p = 0.05, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Depression Severity Measured by PHQ-9
Description: as for outcome 4
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 153 | 132
units on a scale | 5.44 (5.24) | 4.19 (4.51)
Statistical Analysis 1: Comparison: Usual Care-Chronic Disease Management vs P2E2T2 Program; Test type: Equivalence — See Statistical Analysis; p = 0.05, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Depression Severity Measured by PHQ-9
Description: as for outcome 4
Time Frame: 9-months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 149 | 131
units on a scale | 5.69 (6.58) | 4.81 (5.26)
Statistical Analysis 1: Comparison: Usual Care-Chronic Disease Management vs P2E2T2 Program; Test type: Equivalence — See Statistical Analysis; p = 0.05, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Perceived Stress Measured by PSS
Description: Perceived Stress Score (PSS): This is a 4-item instrument administered to patients to measure the degree to which situations in one's life are determined as stressful. The sum total of the responses can range from 0 to 16, with higher scores indicating greater stress. This instrument has acceptable reliability with an alpha of 0.60. This scale has been used and validated in a number of chronic diseases including diabetes.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 155 | 132
units on a scale | 4.98 (3.08) | 5.24 (2.99)
Statistical Analysis 1: Comparison: Usual Care-Chronic Disease Management vs P2E2T2 Program; Test type: Equivalence — See Statistical Analysis; p = 0.05, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Perceived Stress Measured by PSS
Description: as for outcome 7
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 153 | 132
units on a scale | 4.98 (2.99) | 4.64 (3.05)
Statistical Analysis 1: Comparison: Usual Care-Chronic Disease Management vs P2E2T2 Program; Test type: Equivalence — Information in Statistical Analysis; p = 0.05, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Perceived Stress Measured by PSS
Description: as for outcome 7
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 149 | 131
units on a scale | 5.37 (3.48) | 5.22 (3.05)
Statistical Analysis 1: Comparison: Usual Care-Chronic Disease Management vs P2E2T2 Program; Test type: Equivalence — Information included in Statistical Analysis; p = 0.05, Wilcoxon (Mann-Whitney)

10. Other Pre Specified Outcome: PROMIS Emotional Distress Anxiety
Description: PROMIS Emotional Distress Anxiety (www.healthmeasures.net) The Patient Reported Outcomes Measurement Information System Measures (PROMIS) Emotional Distress Anxiety instrument measures self-reported fear, anxious misery and hyperarousal symptoms. Anxiety is best differentiated by symptoms that reflect autonomic arousal and experience of threat. The four-item instrument assesses anxiety over the past seven days using a five item Likert scale (1= not at all, 5 = very much), yielding possible raw scores of 4 to 20. The raw score is translated to a T-score using a score conversion table, with a possible range of 40.3 to 81.6. A score of 50 equals the mean. Higher scores indicate greater emotional distress anxiety. This instrument has demonstrated validity and reliability with an alpha of 0.92 when evaluated in 961 in patients with chronic hepatitis C.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Usual Care-Chronic Disease Management: Usual Care through Chronic Disease Management: The role of the care coordinator is to assess needs of the patient and coordinate healthcare referrals and appointments for the patient, facilitate communication among members of the healthcare team, identify health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient. C
  Usual Care: This program is a well-established program within the UC Davis Health System, providing care coordination to individuals with chronic conditions. Patients can self-refer or are referred by their providers for this service. The role of the care coordinator is to assess needs of the patient and coordinate healthcare referrals and appointments for the patient, facilitate communication among members of the healthcare team, identify health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient.
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 155 | 132
T-score | 51.96 (9.98) | 53.05 (10.10)

11. Other Pre Specified Outcome: PROMIS Emotional Distress Anxiety
Description: PROMIS Emotional Distress Anxiety (www.healthmeasures.net) The Patient Reported Outcomes Measurement Information System Measures (PROMIS) Emotional Distress Anxiety instrument measures self-reported fear, anxious misery and hyperarousal symptoms. Anxiety is best differentiated by symptoms that reflect autonomic arousal and experience of threat. The four-item instrument assesses anxiety over the past seven days using a five item Likert scale (1= not at all, 5 = very much), yielding possible raw scores of 4 to 20. The raw scores are translated to T-scores using a score conversion table, with a possible range of 40.3 to 81.6. A score of 50 equals the mean. Higher scores indicate greater emotional distress anxiety. This instrument has demonstrated validity and reliability with an alpha of 0.92 when evaluated in 961 in patients with chronic hepatitis C.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Usual Care-Chronic Disease Management: Usual Care through Chronic Disease Management: The role of the care coordinator is to assess needs of the patient and coordinate healthcare referrals and appointments for the patient, facilitate communication among members of the healthcare team, identify health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient.
  Usual Care: This program is a well-established program within the UC Davis Health System, providing care coordination to individuals with chronic conditions. Patients can self-refer or are referred by their providers for this service. The role of the care coordinator is to assess needs of the patient and coordinate healthcare referrals and appointments for the patient, facilitate communication among members of the healthcare team, identify health goals in collaboration with the patient and assist them in meeting those goals if requested by the patient. Contact is variable and conducted on a case by case basis.
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 153 | 132
T-score | 49.10 (9.58) | 49.39 (8.88)

12. Other Pre Specified Outcome: PROMIS Emotional Distress Anxiety
Description: as for outcome 11
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 149 | 131
T-score | 51.46 (9.00) | 52.89 (10.64)

13. Other Pre Specified Outcome: PROMIS Physical Function
Description: PROMIS Physical Function (www.healthmeasures.net) The Patient Reported Outcomes Measurement Information System Measures (PROMIS) Physical Function instrument assess the current physical function in the individual. It is a four-item scale measuring self-reported capability of physical activities, using a five item Likert scale (1= not at all, 5 = very much), yielding possible raw scores of 4 to 20. The raw scores are translated to T-scores using a score conversion table, with a possible range of 22.5 to 57.0. A score of 50 equals the mean. Higher scores are associated with higher capability. This instrument has demonstrated validity and reliability with an alpha of 0.91 when evaluated in 4880 patients in a diverse cohort of cancer patients in the US.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 155 | 132
T-score | 30.09 (8.04) | 29.23 (6.01)

14. Other Pre Specified Outcome: PROMIS Physical Function
Description: as for outcome 13
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 153 | 132
T-score | 29.79 (7.51) | 26.26 (6.56)

15. Other Pre Specified Outcome: PROMIS Physical Function
Description: as for outcome 13
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
Number analyzed (Participants) | 149 | 131
T-score | 29.34 (8.27) | 29.77 (7.28)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year
Description: Adverse events that are not Serious Adverse Events were monitored by participant self-report
Arm/Group | Usual Care-Chronic Disease Management | P2E2T2 Program
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/132
Other Adverse Events (participants affected / at risk) | 0/155 | 0/132

LIMITATIONS AND CAVEATS:
Participants might have been more ready to change and to use technology than the general population. With the short intervention, we did not expect change in body mass index or A1C; instead focusing on outcomes important to patients with diabetes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-01-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT02672176/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02672176/SAP_001.pdf